CLINICAL TRIAL: NCT04887454
Title: Optimal Frequency of High-Intensity Interval Training for Centrally Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate Professor and Division Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1v3HIIT
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Obesity; Central Obesity; High-Intensity Interval Training; Aerobic Exercise; Adults; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Once-Weekly HIIT (Experimental): Once-weekly HIIT for 16 weeks, led by certified athletic coaches
  Interventions: Behavioral: Once-Weekly HIIT
- Thrice-Weekly HIIT (Experimental): Thrice-weekly HIIT for 16 weeks, led by certified athletic coaches
  Interventions: Behavioral: Thrice-Weekly HIIT
- Usual Care (Other): Bi-weekly health education, led by research personnel
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Once-Weekly HIIT — Participants in this group will receive a 16-week intervention of HIIT once weekly supervised by certified athletic coaches. Participants will perform four 4-minute intervals at 85%-95% peak heart rate with a 3-minute active recovery between each 4-minute interval. Participants will repeat the 25-minute HIIT bout three times with 30-60 minutes break in between each 25-minute HIIT bout. Health information provided to the usual care control group will be made available to the participants in the HIIT groups.
  Arms: Once-Weekly HIIT
Behavioral: Thrice-Weekly HIIT — Participants in this group will receive a 16-week intervention of HIIT thrice weekly supervised by certified athletic coaches. Participants will perform four 4-minute intervals at 85%-95% peak heart rate with a 3-minute active recovery between each 4-minute interval. Health information provided to the usual care control group will be made available to the participants in the HIIT groups.
  Arms: Thrice-Weekly HIIT
Other: Usual Care — Participants in the usual care control group will receive health education delivered by research personnel. This program will consist of eight two-hour bi-weekly sessions covering major health issues relating to obesity including causes, prevalence, epidemiology, associated diseases, healthy diet, caloric restriction advice, physical activity, stress management, adequate sleep, as well as lifestyle counseling/consultation and goal-setting/record-keeping strategies for behavioral changes.
  Arms: Usual Care

SUMMARY:
The aim of this study is to examine the therapeutic effectiveness of two different exercise frequencies of high-intensity interval training (HIIT; once versus thrice weekly, with matched weekly exercise volume) on improving cardiometabolic risk factors in centrally obese adults.

DETAILED DESCRIPTION:
HIIT is an emerging, popular, promising, cost-effective, and time-efficient exercise modality for managing obesity. Although lower-frequency HIIT is favorable for intervention adherence, the optimal exercise frequency of HIIT for alleviating obesity is unknown.

This study is a three-arm randomized controlled trial. Centrally obese adults will be randomly allocated to three groups: the usual care control, once and thrice-weekly HIIT groups. Led by research personnel, the usual care group will receive obesity-related health education. Led by athletic coaches, the HIIT intervention groups will receive 16 weeks of once or thrice weekly HIIT (with matched weekly exercise volume). Outcome measures of this study will be examined at baseline, 4 months (post-intervention), and 8 months (follow-up), by assessors blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years
* Ethnic Chinese
* Overweight (BMI ≥23 for Asian)
* Centrally obese according to IDF and NCEP with Asian-specific cut-off (waist circumference ≥90 cm for males; ≥80 cm for females)
* Males and females

Exclusion Criteria:

* Medical and somatic conditions that prevent brisk walking
* Chronic diseases affecting mobility and motor function (e.g., neurological disease, musculoskeletal disorder, spinal cord injury, autoimmune, arthritis, Parkinson's Disease)
* Chronic diseases affecting cardiorespiratory and metabolic health (e.g., cancers, cardio-/cerebrovascular diseases, heart disease, diabetes mellitus, pneumonia, chronic pulmonary diseases, nephritis, nephrosis)
* Signs of cardiac arrhythmia indicated by aberrant electrocardiography during incremental VO2max test
* Regular moderate-to-vigorous intensity exercise (≥150 min weekly) in the past 3 months, as screened by a specially designed questionnaire
* Daily smoking habit
* Excess alcohol consumption (daily ≥30g for men, ≥20g for women) in the past six months
* Claustrophobia
* Surgery, therapy or medication for obesity or weight loss in the past six months (e.g., gastric bypass, gastric band, sleeve gastrectomy, gastric reduction duodenal switch, and dietitian-prescribed dietary program)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2024-09-07 (Actual)

PRIMARY OUTCOMES:
Change in Body Fat | Baseline and 4 months
  Total body fat mass will be assessed using dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Change in Body Fat | Baseline and 8 months
  Total body fat mass will be assessed using dual-energy X-ray absorptiometry (DXA)
Change in Abdominal Visceral Fat | Baseline and 4 and 8 months
  Abdominal visceral fat will be assessed using magnetic resonance imaging (MRI)
Change in Abdominal Subcutaneous Fat | Baseline and 4 and 8 months
  Abdominal subcutaneous fat will be assessed using magnetic resonance imaging (MRI)
Change in Body Mass Index | Baseline and 4 and 8 months
  Weight and height will be assessed using a calibrated electronic digital weighing scale and stadiometer respectively
Change in Waist Circumference | Baseline and 4 and 8 months
  Waist circumference will be assessed using an inelastic measuring tape to the nearest 0.1cm on bare skin
Change in Systolic Blood Pressure | Baseline and 4 and 8 months
  Resting systolic blood pressure will be assessed
Change in Diastolic Blood Pressure | Baseline and 4 and 8 months
  Resting diastolic blood pressure will be assessed
Change in Fasting Glucose | Baseline and 4 and 8 months
  Fasting glucose will be analyzed from venous blood by an accredited medical laboratory
Change in Fasting Triglycerides | Baseline and 4 and 8 months
  Fasting triglycerides will be analyzed from venous blood by an accredited medical laboratory
Change in Fasting Low Density Lipoprotein Cholesterol (LDL-C) | Baseline and 4 and 8 months
  Fasting LDL-C will be analyzed from venous blood by an accredited medical laboratory
Change in Fasting High Density Lipoprotein Cholesterol (HDL-C) | Baseline and 4 and 8 months
  Fasting HDL-C will be analyzed from venous blood by an accredited medical laboratory
Change in Fasting Total Cholesterol | Baseline and 4 and 8 months
  Fasting total cholesterol will be analyzed from venous blood by an accredited medical laboratory
Change in Proportion of Metabolic Syndrome Diagnosis | Baseline and 4 and 8 months
  Metabolic syndrome diagnosis will be evaluated with waist circumference, triglycerides, HDL-C, blood pressure, and fasting glucose
Number of Adverse Events | Baseline and 4 and 8 months
  Adverse events related or unrelated to training will be assessed
Change in Organ Fat | Baseline and 4 and 8 months
  Organ fat will be assessed using magnetic resonance imaging (MRI)
Change in SF-12 Physical Component Summary Score | Baseline and 4 and 8 months
  Physical health-related quality of life will be assessed using the Physical Component Summary Score of the 12-Item Short-Form Health Survey (SF-12)
Change in SF-12 Mental Component Summary Score | Baseline and 4 and 8 months
  Mental health-related quality of life will be assessed using the Mental Component Summary Score of the 12-Item Short-Form Health Survey (SF-12)
Change in HADS-D Score | Baseline and 4 and 8 months
  HADS-D score will be assessed using the Depression subscale of the Hospital Anxiety and Depression Scale (HADS-D)
Change in PHQ-9 Score | Baseline and 4 and 8 months
  PHQ-9 score will be assessed using the Patient Health Questionnaire-9 (PHQ-9)
Change in HADS-A Score | Baseline and 4 and 8 months
  HADS-A score will be assessed using the Anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A)
Change in GAD-7 Score | Baseline and 4 and 8 months
  GAD-7 score will be assessed using the General Anxiety Disorder-7 (GAD-7) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Parco M. Siu, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- LKS Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years following the publication of the article.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.

REFERENCES:
- [Derived] Siu PM, Leung CK, Bernal JDK, Yu AP, Recchia F, Tam BT, Fong DYT, Chan DKC, Ngai HH, Lee CH, Yung PSH, Wong SHS, Gibala M. Once and thrice weekly interval training in adults with central obesity: a randomized controlled trial. Nat Commun. 2026 Jan 10;17(1):1410. doi: 10.1038/s41467-025-68149-7. PMID 41519797
- [Derived] Leung CK, Bernal JDK, Yu AP, Recchia F, Tam BT, Fong DYT, Chan DKC, Ngai HH, Lee CH, Yung PSH, Wong SHS, Gibala M, Siu PM. Effects of volume-matched once-weekly and thrice-weekly high-intensity interval training (HIIT) on body adiposity in adults with central obesity: Study protocol for a randomized controlled trial. J Exerc Sci Fit. 2024 Oct;22(4):329-340. doi: 10.1016/j.jesf.2024.05.001. Epub 2024 Jun 14. PMID 38993983